CLINICAL TRIAL: NCT07224282
Title: The Effects of R-1,3-Butanediol With Carbohydrate Supplementation on Cycling Performance Above Lactate Threshold
Brief Title: The Effects of Ketone Supplements With Carbohydrates on Cycling Performance Above Lactate Threshold
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18836
Record Dates: First submitted 2025-10-28; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Exogenous Ketosis
Keywords: Exogenous ketones; Time to fatigue
MeSH Terms: interventions — Carbohydrates; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketone supplementation with carbohydrates (Experimental)
  Interventions: Dietary Supplement: Ketone supplementation; Dietary Supplement: Carbohydrate
- Carbohydrate supplement only (Placebo Comparator)
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Dietary Supplement: Ketone supplementation — 30-gram carbohydrate beverage with 5 grams of R-1,3-Butanediol every 30 minutes of experimental visit
  Arms: Ketone supplementation with carbohydrates
Dietary Supplement: Carbohydrate — 30-gram carbohydrate beverage with bitter flavoring
  Other Names: Dextrose

SUMMARY:
The goal of this clinical trial is to determine whether a ketone supplement with carbohydrates extends time to fatigue during cycling compared with a carbohydrate-only supplement in healthy, trained cyclists aged 18-55. The main questions it aims to answer are:

Is the time to fatigue increased with ketone supplementation and carbohydrates compared to carbohydrates alone? Will ketone supplementation with carbohydrates produce lower blood lactate concentrations compared to carbohydrates alone?

Participants will:

* Perform a staged maximal cycling exercise test on a stationary bicycle.
* Finger prick to obtain a drop of blood for lactate measurements.
* Wear a mask connected to a metabolic cart to measure breath contents.
* Perform a cycling exercise test to fatigue for at least one hour.
* Consume either a ketone supplement with carbohydrates or a carbohydrate supplement during the exercise at least 4 times.
* Finger prick to obtain a drop of blood to measure blood lactate, ketones, and glucose.

DETAILED DESCRIPTION:
The significance of this study is to address gaps in the literature by investigating the combined effects of R-1,3-Butanediol and carbohydrate supplementation on cycling performance during steady-state exercise above the lactate threshold. Participants include:

1. Trained cyclists ages 18-55

   1. ≥ 6 hours of cycle training per week.
   2. Above average VO2max for their age range per ACSM guidelines.
2. The sample is drawn from the University of Oklahoma, local cycling events in Oklahoma, and local bicycle shops.

There will be a total of three visits, lasting approximately one hour and separated by at least 7 days. The protocol begins with a familiarization visit, during which participants complete a maximal graded exercise test. They are instructed to be at least 4 hours postabsorptive and not complete strenuous exercise within 24 hours of the initial visit, and each participant signs an informed consent form, fills out a POMS questionnaire, and exercise history questionnaire (PAR-Q). Participants' height and weight were recorded, and their bicycles will be connected to the cycling trainer or will use the Zwift One stationary bicycle. To determine VO2 max and lactate threshold, a continuous incremental cycling test will be performed. The test begins at 1 watt per kilogram of body weight and increases 0.5 watts per kilogram of body weight every 3 minutes until two of the following were reached: volitional fatigue, inability to maintain cadence within 10 rpm of their preferred cadence, maximal heart rate within 10 bpm of age-predicted max heart rate, or respiratory exchange ratio greater than 1.10 The intent is to provide insights into metabolic and performance responses beyond traditional exercise intensities. The findings could inform endurance athletes and coaches on nutritional strategies for sustaining performance during high-intensity efforts.The study aims to investigate the performance effects of a ketone supplement (R-1,3-Butanediol) with carbohydrate supplementation on cycling performance above the lactate threshold. It aims to determine whether time to fatigue will be affected and if blood lactate concentrations will decrease due to ketone supplementation. Hypotheses include:

Time to fatigue is increased with ketone supplementation and carbohydrates compared to carbohydrates alone.

Ketone supplementation with carbohydrates will produce lower blood lactate concentrations compared to carbohydrates alone.

ELIGIBILITY:
Inclusion Criteria:

* Highly trained males and females
* Ages 18-55
* Greater than or equal to six hours of cycling training per week
* Participants from the University of Oklahoma, Oklahoma cycling teams, and local cycling races in Oklahoma.

Exclusion Criteria:

* Cardiovascular disease
* Respiratory disease
* Gastrointestinal disease
* Metabolic disease
* Kidney disease
* Neurological disease
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Time to fatigue | Through study completion, an average of 2 weeks.

SECONDARY OUTCOMES:
Blood lactate | Through study completion, an average of 2 weeks.
Blood Glucose | Through study completion, an average of 2 weeks.
Beta-hydroxybutyrate levels | Through study completion, an average of 2 weeks.
  Using a finger prick to obtain a drop of blood to measure beta-hydroxybutyrate levels in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma, Norman, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltz NM, Gibson AL, Janot JM, Kravitz L, Mermier CM, Dalleck LC. Graded Exercise Testing Protocols for the Determination of VO2max: Historical Perspectives, Progress, and Future Considerations. J Sports Med (Hindawi Publ Corp). 2016;2016:3968393. doi: 10.1155/2016/3968393. Epub 2016 Dec 25. PMID 28116349
- [Background] Dearlove DJ, Harrison OK, Hodson L, Jefferson A, Clarke K, Cox PJ. The Effect of Blood Ketone Concentration and Exercise Intensity on Exogenous Ketone Oxidation Rates in Athletes. Med Sci Sports Exerc. 2021 Mar 1;53(3):505-516. doi: 10.1249/MSS.0000000000002502. PMID 32868580
- [Background] Leckey JJ, Ross ML, Quod M, Hawley JA, Burke LM. Ketone Diester Ingestion Impairs Time-Trial Performance in Professional Cyclists. Front Physiol. 2017 Oct 23;8:806. doi: 10.3389/fphys.2017.00806. eCollection 2017. PMID 29109686
- [Background] Shaw DM, Merien F, Braakhuis A, Plews D, Laursen P, Dulson DK. The Effect of 1,3-Butanediol on Cycling Time-Trial Performance. Int J Sport Nutr Exerc Metab. 2019 Sep 1;29(5):466-473. doi: 10.1123/ijsnem.2018-0284. PMID 30632425
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046